CLINICAL TRIAL: NCT03407547
Title: Neural Correlates of Upper Limb Somatosensory Impairments and Recovery in the Acute Phase After Stroke: an EEG Investigation
Brief Title: A Study Exploring Brain Activity in Relation to Sensory Arm Impairments in the Early Stages of Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S61174
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: upper limb; recovery; somatosensory; impairment; electroencephalography; acute phase
MeSH Terms: conditions — Stroke | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electroencephalography — EEG is a device to measure brain activity via surface electrodes

SUMMARY:
This clinical study is organized for people with stroke often experience difficulties with their sensation in their upper limb. New technologies may be able to help these important problems. However, there is currently not enough knowledge about how the brain recovers in people with sensory impairments in their arm and hand. Using a non-invasive technique of recording brain activity, known as electroencephalography (EEG), brain activity in combination with somatosensation of the hand will be measured. Therefore, the purpose of this study will be to analyse brain activity in relation to somatosensory impairments after stroke during the first two weeks after stroke.

ELIGIBILITY:
Participants will be recruited during the first 2-3 days post-stroke. They should have:

1. a first-ever unilateral, supra-tentorial stroke, as defined by Wold Health Organisation;
2. admission to the acute hospital,
3. deficit in distal pinprick somatosensory measured by Rivermead assessment of somatosensory performance (score of ≤4) and/or motor impairment measured by Fugl Meyer Assessment (score of ≤12 out of 14),
4. the age of > 18 years and
5. the ability to provide informed consent.

Healthy adults will also be recruited and they should have:

1. no history of sensory impairments in their hands
2. the age of > 18 years and
3. the ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensory Evoked Potential Latency | First 2 weeks post-stroke
  EEG measurement
Sensory Evoked Potential Amplitude | First 2 weeks post-stroke
  EEG measurement

SECONDARY OUTCOMES:
Fugl Meyer Assessment | First 2 weeks post-stroke
  Upper limb motor impairment measurement
Wolf Motor Function Test | First 2 weeks post-stroke
  Upper limb activities measurement
Perceptual Threshold of Touch | First 2 weeks post-stroke
  Light touch of the palmar surface of index finger
Erasmus modified Nottingham Sensory Assessment | First 2 weeks post-stroke
  Measures somatosensation of the upper limb and hand
Nottingham Sensory Assessment | First 2 weeks post-stroke
  Measures stereognosis
Montreal Cognitive Assessment | First 2 weeks post-stroke
  Measures cognition

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luc Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No